CLINICAL TRIAL: NCT01768078
Title: Interest of Intravitreal Corticotherapy as the First-line Treatment for Post-operative Endophthalmitis.
Acronym: Endophtalmitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Creuzot-Garcher PHRC IR 2007
Record Dates: First submitted 2013-01-08; First posted 2013-01-15 (Estimated); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Post-operative Endophthalmitis
MeSH Terms: interventions — Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- with corticoids (Experimental)
  Interventions: Procedure: Intravitreal injection of Betamethasone + antibiotics
- without corticoids (Other)
  Interventions: Procedure: Intravitreal injection of antibiotics

INTERVENTIONS:
Procedure: Intravitreal injection of Betamethasone + antibiotics
  Arms: with corticoids
Procedure: Intravitreal injection of antibiotics
  Arms: without corticoids

SUMMARY:
One useful effect of early intravitreal corticotherapy is to diminish inflammatory complications after endophthalmitis, which may cause, at least in part, serious complications (retinal detachment, macular edema) which are, more than the infection, causes of the complications seen after acute endophthalmitis.

ELIGIBILITY:
Inclusion Criteria:

* All patients male or female with no age limit
* Hospitalized for the diagnosis and treatment of acute endophthalmitis following cataract surgery
* Who had given their consent after being informed about intravitreal corticotherapy

Exclusion Criteria:

* Patients who refused or were unable to give their consent
* Prior intravitreal corticotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Measure the evolution of visual acuity | up to12 months

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CHU de Besançon, Besançon
  - CHU, Dijon
  - CHU de Grenoble, Grenoble
  - CHU de Nancy, Nancy
  - CHU de Saint Etienne, Saint-Etienne
  - CHU de Strasbourg, Strasbourg